CLINICAL TRIAL: NCT02740868
Title: Development of Hyperpolarized Xenon-129 and Inert Fluorinated Gas Lung Magnetic Resonance Imaging: Comparative Pilot Study of Healthy Volunteers and Participants With Pulmonary Disease
Brief Title: Xenon-129 and Inert Fluorinated Gas Lung Magnetic Resonance Imaging: Study of Healthy Volunteers and Participants With Pulmonary Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Giles Santyr, Senior Scientist, The Hospital for Sick Children
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1000048243
Record Dates: First submitted 2015-08-19; First posted 2016-04-15 (Estimated); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Cystic Fibrosis; Asthma
Keywords: Magnetic Resonance Imaging,cystic fibrosis,asthma,healthy
MeSH Terms: conditions — Cystic Fibrosis; Asthma | interventions — Xenon-129; perflutren; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy (Active Comparator): Healthy Participants ages 8 and older. Participants with inhale hyperpolarized xenon-129 which is used as a contrast agent for lung imaging. Perfluoropropane will also be used as a contrast agent for MRI. Perfluoropropane will be inhaled as a normoxic mixture (21% O2 and 79% perfluoropropane). Participants will undergo magnetic resonance imaging and lung clearance index.
  Interventions: Drug: Xenon-129 and Perfluoropropane (19F); Device: Magnetic Resonance Imaging; Device: Lung Clearance Index
- Cystic Fibrisos (Active Comparator): Participants with cystic fibrosis ages 8 and older.Participants with inhale hyperpolarized xenon-129 which is used as a contrast agent for lung imaging. Perfluoropropane will also be used as a contrast agent for MRI. Perfluoropropane will be inhaled as a normoxic mixture (21% O2 and 79% perfluoropropane). Participants will undergo magnetic resonance imaging and lung clearance index.
  Interventions: Drug: Xenon-129 and Perfluoropropane (19F); Device: Magnetic Resonance Imaging; Device: Lung Clearance Index
- Asthma (Active Comparator): Participants with asthma ages 8 and older.Participants with inhale hyperpolarized xenon-129 which is used as a contrast agent for lung imaging. Perfluoropropane will also be used as a contrast agent for MRI. Perfluoropropane will be inhaled as a normoxic mixture (21% O2 and 79% perfluoropropane). Participants will undergo magnetic resonance imaging and lung clearance index.
  Interventions: Drug: Xenon-129 and Perfluoropropane (19F); Device: Magnetic Resonance Imaging; Device: Lung Clearance Index

INTERVENTIONS:
Drug: Xenon-129 and Perfluoropropane (19F) — Xenon gas and perfluoropropane to be inhaled by research participants
  Other Names: 129Xe and 19F
Device: Magnetic Resonance Imaging — Lung imaging will be performed for participants using MRI for all 3 arms
  Other Names: MRI
Device: Lung Clearance Index — Lung clearance index (measure of lung health) will be performed for all participants of all 3 arms
  Other Names: LCI

SUMMARY:
Aim of this study is to evaluate image quality and reproducibility of Xenon-129 and Inert fluorinated (19F) gas Magnetic Resonance Imaging (MRI) and to evaluate changes in lung structure and function in participants with cystic fibrosis (CF) and asthma compared to healthy controls.

DETAILED DESCRIPTION:
Hyperpolarized noble gas magnetic resonance (MR) lung imaging is a relatively new imaging method that allows depiction of both lung function and morphology. Hyperpolarized gases are a new class of MR contrast agent which, when inhaled, provide high temporal and spatial resolution MR images of the lung airspaces. Since no ionizing radiation is involved, hyperpolarized gas MR imaging is ideal for the evaluation of lung diseases especially in children. With hyperpolarized gases, the nuclear spins of the gas atoms are brought into alignment outside of the MR scanner via a process called optical pumping; this yields high polarizations and permits visualization of the lung airspaces with MR imaging (despite the low physical density of the gas in the lung). Two non-radioactive (i.e. stable) isotopes of noble gases helium-3 and xenon-129 can be hyperpolarized. Until recently, higher polarizations could be achieved with helium-3 than with xenon-129, so in humans, helium-3 was more commonly used for hyperpolarized gas MR imaging of the lungs. Recently, the technology has been developed to provide large quantities of highly polarized xenon-129. Helium-3 gas is also extremely expensive and since there are limited reserves of the gas, difficult to procure for research. Unlike helium-3, since xenon-129 is naturally present in the atmosphere, it is less expensive and easier to procure for imaging.

Several applications of xenon-129 MR imaging are under development, including diffusion-weighted and relaxation-weighted imaging. These techniques take advantage of the fact that the rate of loss of xenon-129 polarization is significantly influenced by the local blood flow and concentration of molecular oxygen, as well as the restriction of xenon-129 diffusion by small airway space dimensions. These data can be used to create maps of the lung reflecting regional ventilation/perfusion and micro-airway sizes. Other data that can be obtained with xenon-129 MRI include the volumes of ventilated and unventilated lungs which can subsequently be analyzed to determine the homogeneity of gas distribution within the airspaces. These data can be used to study the structural and functional changes taking place in the lungs associated with pulmonary diseases like CF and asthma. It might provide a diagnostic tool that is able to detect pulmonary diseases more sensitively than the current gold standard measurements of spirometry and plethysmography, and thus prevent irreparable and irreversible damage to the lungs in the early stages of disease.

19F MRI is an emergent technology for the imaging of lung ventilation and function. Similar to HP 129Xe MRI, this technique involves the imaging of an inhaled tracer (inert fluorinated gases) to visualize the airspaces of the lungs. Fluorinated gases such as perfluoropropane have been approved for use as an investigational inhaled contrast at several institutions globally, including a Canadian institution in Thunder Bay, Ontario. Fluorinated gases are non-toxic, commercially available, relatively inexpensive, and have favourable physical/magnetic properties for MRI17-20. Most importantly, unlike 129Xe MRI, fluorinated gases do not require hyperpolarization prior to imaging to boost detectable signal, instead relying on a relatively high number of 19F atoms per molecule and rapid, repeated imaging to enable sufficient signal averaging3. This is a significant advantage compared to HP 129Xe MRI which requires special polarizing equipment; a major barrier to widespread implementation. Despite this, the achievable image quality is generally poorer than 129Xe MRI. Nevertheless, recent improvements in hardware, software and fluorinated gases may enable 19F MRI to provide similar and/or complimentary information compared to HP 129Xe MRI at lower cost and with reduced requirements for hardware and infrastructure21.

Additionally, the paramagnetism of molecular oxygen (O2), which detrimentally impacts the hyperpolarization of 129Xe, does not significantly impact inert fluorinated gases. Therefore, these gases may be prepared in normoxic mixtures prior to administration to participants, rather than in anoxic mixtures as is typically done with 129Xe. This, alongside the fact that irreversible loss of magnetization is not a concern with fluorinated gases, presents the opportunity to perform free-breathing, extended imaging of the lungs. Imaging data acquired during free-breathing can potentially resolve gas kinetics (i.e., gas-wash-in, wash-out, and fractional ventilation)22,23 in a manner that is more feasible and tolerable than with HP noble gases.

Due to the lack of studies evaluating 19F MRI in pediatric lung disease, in this study we aim to develop and test necessary hardware/software for 19F MRI of the lungs children with and without history of respiratory disease and compare to HP 129Xe MRI.

ELIGIBILITY:
Inclusion Criteria:

1. Participants male and female aged 8 years old and older.
2. Participants have no smoking history.
3. For participants with CF and asthma, a clinical diagnosis is necessary and they should be at their baseline level of symptom control based on history.
4. Participants should have a FEV1%pred value greater than 40%.
5. Participant understands the study procedures and is willing to participate in the study as indicated by signature on the informed consent or assent.
6. Participant must be able to perform a breath hold for 20s or less.
7. Participant able to perform reproducible pulmonary function tests (i.e., the 3 best acceptable spirograms have FEV1 values that do not vary more than 5% of the largest value or more than 100 ml, whichever is greater).

For the PEx sub-cohort, admission to the Hospital for Sick Children for a pulmonary exacerbation (based on clinical or pulmonary function assessment). Children who will be admitted and then discharged on home IV antibiotics may also be included in this study.

Exclusion Criteria:

1. Participant is, in the opinion of the investigator, mentally or legally incapacitated, preventing informed consent/assent from being obtained, or cannot read or understand the written material.
2. Participant has a history of cardiovascular disorders including coronary insufficiency, cardiac arrhythmias, severe hypertension.
3. Other than for the PEx sub-cohort, participant has had a cold or respiratory infection in the last four weeks.
4. Participant requires supplemental oxygen or has a daytime room air oxygen saturation ≤ 95%.
5. Participant is unable to perform spirometry or plethysmography maneuvers.
6. Participant is pregnant or lactating.
7. In the investigator's opinion, participant suffers from any physical, psychological or other condition(s) that might prevent performance of the MRI, such as severe claustrophobia.
8. Participant has an MRI incompatible device or any metal in their body which cannot be removed, including but not limited to pacemakers, neurostimulators, biostimulators, implanted insulin pumps, aneurysm clips, bio prosthetic, artificial limb, metallic fragment or foreign body, shunt, surgical staples (including clips or metallic sutures and/or ear implants).

   -

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-08; Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Significant differences in lung function between CF and healthy group and asthma and healthy group for ventilation defect percent (VDP) measurement | 1 year
  To evaluate image quality and reproducibility of 129Xe and inert fluorinated (19F) gas MRI and to evaluate changes in lung structure and function in participants with cystic fibrosis (CF) and asthma compared to healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Giles Santyr, PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Munidasa S, Couch MJ, Rayment JH, Voskrebenzev A, Seethamraju R, Vogel-Claussen J, Ratjen F, Santyr G. Free-breathing MRI for monitoring ventilation changes following antibiotic treatment of pulmonary exacerbations in paediatric cystic fibrosis. Eur Respir J. 2021 Apr 15;57(4):2003104. doi: 10.1183/13993003.03104-2020. Print 2021 Apr. No abstract available. PMID 33303537
- [Derived] Kanhere N, Couch MJ, Kowalik K, Zanette B, Rayment JH, Manson D, Subbarao P, Ratjen F, Santyr G. Correlation of Lung Clearance Index with Hyperpolarized 129Xe Magnetic Resonance Imaging in Pediatric Subjects with Cystic Fibrosis. Am J Respir Crit Care Med. 2017 Oct 15;196(8):1073-1075. doi: 10.1164/rccm.201611-2228LE. No abstract available. PMID 28245140